CLINICAL TRIAL: NCT05671510
Title: Phase 3, Two-stage, Randomized Study of ONC-392 Versus Docetaxel in Metastatic Non-Small Cell Lung Cancers That Progressed on PD-1/PD-L1 Inhibitors
Brief Title: ONC-392 Versus Docetaxel in Metastatic NSCLC That Progressed on PD-1/PD-L1 Inhibitors
Acronym: PRESERVE-003
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: OncoC4, Inc. (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRESERVE-003
Record Dates: First submitted 2022-12-26; First posted 2023-01-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, active controlled, multi-center Phase 3 study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Gotistobart 6 mg/kg with 2 loading doses of 10 mg/kg, Q3W (Experimental): Gotistobart will be administrated by IV infusion in 60 minutes on day 1 of each cycle. A cycle is 21 days.
  Interventions: Drug: Gotistobart
- Arm 2: Docetaxel 75 mg/m2, Q3W (Active Comparator): Docetaxel will be administrated by IV infusion in 60 minutes on day 1 of each cycle. A cycle is 21 days.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Gotistobart — Gotistobart will be administrated through IV infusion over 60 minutes, once every 21 days in assigned dose.
  Other Names: A humanized anti-CTLA4 IgG1 monoclonal antibody; ONC-392; BNT316
  Arms: Arm 1: Gotistobart 6 mg/kg with 2 loading doses of 10 mg/kg, Q3W
Drug: Docetaxel — Docetaxel will be administrated through IV infusion over 60 minutes, once every 21 days in 75mg/m2 dose.
  Other Names: Docefrez; Taxotere
  Arms: Arm 2: Docetaxel 75 mg/m2, Q3W

SUMMARY:
The goal of this Phase 3 clinical trial is to study the safety and efficacy of the nextgen anti-CTLA-4 antibody, gotistobart (ONC-392/BNT316), in patients with metastatic non-small cell lung cancer who have disease progressed on anti-PD-1/PD-L1 antibody based therapy. The study will test whether gotistobart, in comparison with chemotherapy agent docetaxel, could prolong the life for NSCLC patients. Patients will be randomized to be treated with either gotistobart or docetaxel, IV infusion, once every 21 days, for up to 17 cycles in approximately one year.

DETAILED DESCRIPTION:
This is a seamless 2-stage, randomized, open-label, active-controlled, Phase 3 study. The study population consists of patients with NSCLC who progressed on PD-1/PD-L1 inhibitor. Approximately 630 patients will be enrolled.

Two gotistobart dosing regimens will be tested in Stage I, and one will be selected for Stage II.

Stage I, the dose-confirmation stage, will assess the efficacy and safety of two gotistobart dosing regimens (3 mg/kg Q3W and 6 mg/kg Q3W with 2 loading doses of 10 mg/kg Q3W) in comparison to docetaxel 75 mg/m2 Q3W.

Stage II will assess the safety and efficacy of gotistobart at the selected dosing regimen versus docetaxel on squamous cell NSCLC. Patients will be randomized 1:1 to receive either gotistobart at the selected dosing regimen or docetaxel.

ELIGIBILITY:
Inclusion Criteria (Major criteria):

1. Adult (≥ 18 years), all genders, capable of signing informed consent.
2. Histologically- or cytologically- confirmed diagnosis of metastatic squamous NSCLC, metastasis can be regional lymph nodes or distant organs.
3. Radiographic progression after treatment with the most recent line of treatment being either 3a or 3b:

   1. At least 12 weeks of PD-1/PD-L1 inhibitor in combination with platinum-based chemotherapy;
   2. Prior treatment with at least 2 cycles of a platinum-based chemotherapy, followed by at least 12 weeks of standard doses of PD-1 or PD-L1 inhibitor-based immunotherapy.

   Antibodies against CTLA-4, LAG-3, TIGIT, VEGF or VEGFR in combination with PD-1/PD-L1 inhibitor are allowed.
4. At least one measurable tumor lesion according to RECIST 1.1.
5. ECOG score of 0 or 1.
6. Adequate organ functions. Serum LDH level ≤ 2xULN.
7. Life expectancy ≥ 3 months.

Exclusion Criteria (Major criteria):

1. Cancer treatment related AEs have not recovered to NCI CTCAE grade≤ 1 except endocrinopathy.
2. Last anti-PD-1/PD-L1 dosing within 28 days prior to first dose of study treatment.
3. Receiving systemic steroid therapy with >10 mg/day prednisone or equivalent within 7 days prior to the first dose of study treatment.
4. Having documented actionable mutations or genomic alterations in any of the following genes: EGFR, ALK, ROS1, HER2, MET, BRAF, RET or NTRK;. Exception: KRAS mutations are not excluded.
5. Patients who have symptomatic brain metastasis. Palliative radiotherapy or radiosurgery to brain metastasis within 14 days of the first dose of study drug.
6. Active GI disease, including peptic ulcer disease, pancreatitis, diverticulitis, or inflammatory bowel disease.
7. Active interstitial lung disease (ILD) or non-infectious pneumonitis.
8. Active infections with IV antibiotics within 14 days prior to first dose of study treatment.
9. Impaired heart function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 36 months
  OS is defined as the time from randomization to the date of death by any cause. Kaplan-Meier estimates of median OS time will be presented by treatment arm with two sided 95% CIs.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 36 months
  Objective response rate (ORR) as assessed by the Investigator per RECIST 1.1
Progression-free survival (PFS) | 36 months
  Progression-free survival (PFS) as assessed by Investigator per RECIST 1.1
Treatment emergent adverse events, treatment related adverse events and immune related adverse events. | 36 months
  Incidence of TEAEs, TRAEs, irAEs will be calculated. The AEs leading to treatment discontinuation will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Socinski, MD, Principal Investigator — Advent Health System; Tianhong Li, MD, PhD, Principal Investigator — University of California, Davis; Kai He, MD, PhD, Principal Investigator — Ohio State University
Locations (152):
- United States (46):
  - XCancer/Dothan Hematology & Oncology - 1114, Dothan, Alabama
  - Genesis Cancer and Blood Institute - 1123, Russellville, Arkansas
  - The Oncology Institute (TOI) Clinical Research - 1109, Cerritos, California
  - Emad Ibrahim MD Inc. - 1147, Redlands, California
  - UC Davis Comprehensive Cancer Center - 1103, Sacramento, California
  - Bass Medical Group - 1155, Walnut Creek, California
  - Nuvance Health - 1118, Norwalk, Connecticut
  - D&H Cancer Research Center LLC - 1153, Margate, Florida
  - Ocala Oncology Center PL - 1102, Ocala, Florida
  - AdventHealth Cancer Institute - 1105, Orlando, Florida
  - Orlando Health - 1130, Orlando, Florida
  - Florida Cancer Specialists -South - 1126, Sarasota, Florida
  - Florida Cancer Specialists -North - 1125, The Villages, Florida
  - Florida Cancer Specialists -East - 1124, West Palm Beach, Florida
  - Orchard Healthcare Research, Inc. - 1116, Skokie, Illinois
  - Springfield Clinic - The Cancer Center - 1110, Springfield, Illinois
  - Fort Wayne Medical Oncology - 1133, Fort Wayne, Indiana
  - Deaconess Chancellor Center for Oncology - 1131, Newburgh, Indiana
  - Cotton O'Neil Clinical Research Center - 1151, Topeka, Kansas
  - University of Kentucky - Markey Cancer Center - 1112, Lexington, Kentucky
  - Norton Cancer Institute - 1108, Louisville, Kentucky
  - Jefferson City Medical Group - 1145, Jefferson City, Missouri
  - MidAmerica Cancer Care - 1163, Kansas City, Missouri
  - Astera Cancer Care - 1128, East Brunswick, New Jersey
  - Duke University Medical Center - 1158, Durham, North Carolina
  - Miami Valley Hospital - 1115, Centerville, Ohio
  - University of Cincinnati Cancer Center - 1107, Cincinnati, Ohio
  - The Ohio State University James Cancer Center - 1104, Columbus, Ohio
  - Tri County Hematology & Oncology Associates, Inc - 1156, Massillon, Ohio
  - Oklahoma Cancer Specialists and Research Institute - 1154, Tulsa, Oklahoma
  - Oncology Associates of Oregon - 1138, Eugene, Oregon
  - St. Luke's University Health Network - 1179, Bethlehem, Pennsylvania
  - Donald Guthrie Foundation - 1135, Sayre, Pennsylvania
  - Cancer Care Associates of York, Inc. - 1113, York, Pennsylvania
  - University of Tennessee Medical Center - 1146, Knoxville, Tennessee
  - Sarah Cannon Research Institute - Tennessee Oncology at Nashville - 1119, Nashville, Tennessee
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center (USOR) - 1140, Dallas, Texas
  - Texas Oncology - Denison - 1139, Denison, Texas
  - Oncology Consultants, P.A. - 1120, Houston, Texas
  - Oncology and Hematology of South Texas - 1165, Laredo, Texas
  - Texas Oncology - McAllen - 1132, McAllen, Texas
  - Texas Oncology -San Antonio - 1122, San Antonio, Texas
  - NEXT Oncology - Virginia - 1129, Fairfax, Virginia
  - Virginia Cancer Institute - 1149, Henrico, Virginia
  - Virginia Oncology Associates - 1136, Norfolk, Virginia
  - West Virginia University Cancer Institute - 1172, Morgantown, West Virginia
- Australia (4):
  - Bankstown Hospital - 3305, Bankstown, New South Wales
  - Mater - 3301, Newstead, Queensland
  - Cancer Research SA - 3303, Adelaide, South Australia
  - Western Health - Sunshine Hospital - 3307, St Albans, Victoria
- Belgium (4):
  - AZ Maria Middelares - 2104, Ghent
  - Jessa Ziekenhuis (Jessa Hospital) - Campus Salvator - 2102, Hasselt
  - C. H. R. de la Citadelle - 2103, Liège
  - Vitaz - Sint-niklaas Moerland - 2101, Sint-Niklaas
- Canada (3):
  - BC Cancer Centre - Kelowna - 1203, Kelowna, British Columbia
  - Saskatchewan Cancer Agency - Regina - 1201, Regina, Saskatchewan
  - Saskatchewan Cancer Agency - Saskatoon Cancer Centre - 1202, Saskatoon, Saskatchewan
- China (40):
  - The First Affiliated Hospital of Anhui Medical University - 3221, Hefei, Anhui
  - Anhui Medical University - The Second Hospital - 3222, Hefei, Anhui
  - Beijing Cancer Hospital - 3205, Beijing, Beijing Municipality
  - Cancer Hospital, Chinese Academy of Medical Sciences - 3211, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital - 3225, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University - 3210, Xiamen, Fujian
  - Dongguan People's Hospital - 3206, Dongguan, Guangdong
  - Guangdong Provincial People's Hospital - 3201, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University - 3203, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangdong Pharmaceutical University - 3215, Guangzhou, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region - 3228, Nanning, Guangxi
  - Hainan General Hospital - 3202, Haikou, Hainan
  - Affiliated Hospital of Hebei University - 3214, Zhengzhou, Hebei
  - The Affiliated Tumor Hospital of Harbin Medical University - 3232, Harbin, Heilongjiang
  - Henan Cancer Hospital - 3226, Zhengzhou, Henan
  - The First Affliated Hospital of Zhengzhou University - 3207, Zhengzhou, Henan
  - Renmin Hospital of Wuhan University - 3216, Wuhan, Hubei
  - Union Hospital Tongji Medical College - 3212, Wuhan, Hubei
  - Xiangya Hospital, Central South University - 3223, Changsha, Hunan
  - Hunan Cancer Hospital - 3209, Changsha, Hunan
  - The Second Affiliated Hospital of Soochow University - 3217, Suzhou, Jiangsu
  - Xuzhou Medical University - The Affiliated Hospital - 3234, Xuzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University - 3224, Nanchang, Jiangxi
  - Jinan Central Hospital - 3230, Jinan, Shandong
  - Shanxi Bethune Hospital - 3233, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University - 3218, Xi’an, Shanxi
  - Chengdu Seventh People's Hospital - 3229, Chengdu, Sichuan
  - Sichuan Cancer Hospital - 3227, Chengdu, Sichuan
  - Chongqing University Cancer Hospital - 3213, Chongqing, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital - 3208, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital - 3231, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine - 3219, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine - 3220, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital - 3204, Hangzhou, Zhejiang
  - China-Japan Friendship Hospital - 3236, Beijing
  - West China Hospital, Sichuan University - 3238, Chengdu
  - Nanjing Medical University (NMU) - Nanjing First Hospital - 3239, Jiangse
  - Weifang Second People's Hospital - 3235, Shandong
  - Tongji University - Shanghai Oriental Hospital (Shanghai East Hospital) - 3240, Shanghai
  - Hubei Cancer Hospital - 3237, Wuhan
- Germany (6):
  - Städt. Klinikum München GmbH - 2204, Bogenhausen
  - Kliniken Essen-Mitte - 2206, Essen
  - Klinikum Esslingen GmbH - 2201, Esslingen am Neckar
  - Lungenfachklinik Immenhausen - 2202, Immenhausen
  - Klinikverbund Allgaü - Klinikum Kempten - 2205, Immenstädt
  - Asklepios Fachkliniken Muenchen-Gauting - 2203, Muenchen-Gauting
- Italy (11):
  - Clinica Oncologica Ospedali Riuniti Ancona - 2311, Ancona
  - IRCCS Istituto Tumori Giovanni Paolo II - 2306, Bari
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII - 2310, Bergamo
  - Humanitas Istituto Clinico Catanese - 2312, Catania
  - Ospedale San Raffaele - 2307, Milan
  - Fondazione IRCCS Instituto Tumori Di Milano - 2305, Milan
  - Ospedale San Gerardo di Monza - 2302, Monza
  - Azienda Ospedaliera Universitaria "Federico II" - 2304, Naples
  - AOU Policlinico Giaccone, Università di Palermo - 2309, Palermo
  - Universita degli Studi di Perugia - Ospedale Santa Maria della Misericordia - 2308, Perugia
  - Universita Campus Bio-medico Di Roma (UCBM) - Policlinico Universitario - 2303, Roma
- Netherlands (3):
  - Antoni van Leeuwenhoek - 2703, Amsterdam
  - Rijnstate Ziekenhuis - 2701, Arnhem
  - ETZ Elisabeth - 2704, Tilburg
- South Korea (7):
  - Chungbuk National University Hospital - 3101, Cheongju-si
  - Keimyung University Dongsan Hospital - 3102, Daegu
  - National Cancer Center - 3107, Goyang-si
  - Severance Hospital, Yonsei University Health System - 3104, Seoul
  - Asan Medical Centre - 3103, Seoul
  - Korea University Guro Hospital - 3106, Seoul
  - The Catholic University of Korea, St Vincent's Hospital - 3105, Suwon
- Spain (6):
  - Hospital General Universitario de Elche - 2401, Elche
  - Hospital Universitario Lucus Augusti - 2405, Lugo
  - Hospital General Universitario Gregorio Marañon - 2404, Madrid
  - Hospital Regional Universitario de Malaga - 2403, Málaga
  - Hospital General Universitario de Valencia - 2406, Valencia
  - Fundacion Instituto Valenciano De Oncologia (IVO) - 2402, Valencia
- Turkey (Türkiye) (12):
  - Adana Sehir Hastanesi - 2602, Adana
  - Baskent University Adana - 2601, Adana
  - Hacettepe Universitesi - 2609, Ankara
  - Ankara Bilkent Sehir Hastanesi - 2610, Ankara
  - Akdeniz University Medical Hospital - 2606, Antalya
  - Trakya University Faculty of Medicine Edirne - 2608, Edirne
  - Istanbul Üniversitesi Onkoloji Enstitüsü - 2613, Fatih
  - Koc Universitesi - 2611, Istanbul
  - Göztepe Prof Dr. Suleyman Yalcin City Hospital - 2605, Istanbul
  - Istanbul Bakirkoy Sadi Konuk - 2604, Istanbul
  - Medipol University Medical Faculty Hospital - 2603, Istanbul
  - Izmir Ekonomi Universitesi Medical Point Hastanesi - 2607, Izmir
- United Kingdom (10):
  - University Hospital Birmingham (UHB) / Queen Elizabeth Hospital Birmingham - 2801, Birmingham, England
  - Cambridge University Hospitals - 2804, Cambridge, England
  - Royal Devon University Healthcare NHS - 2808, Exeter, England
  - University Hospital Leicester - 2806, Leicester, England
  - Barts Health NHS Trust (St. Bartholomew's Hospital) - 2803, London, England
  - South Tees Hospitals - 2807, Middlesbrough, England
  - Torbay and South Devon NHS Foundation Trust - 2805, Torquay, England
  - The Christie NHS Foundation Trust - 2802, Manchester, London
  - Edinburgh Cancer Centre - 2809, Edinburgh, Scotland
  - University College London Hospital - 2811, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Y, Du X, Liu M, Tang F, Zhang P, Ai C, Fields JK, Sundberg EJ, Latinovic OS, Devenport M, Zheng P, Liu Y. Hijacking antibody-induced CTLA-4 lysosomal degradation for safer and more effective cancer immunotherapy. Cell Res. 2019 Aug;29(8):609-627. doi: 10.1038/s41422-019-0184-1. Epub 2019 Jul 2. PMID 31267017
- [Background] Liu Y, Zheng P. Preserving the CTLA-4 Checkpoint for Safer and More Effective Cancer Immunotherapy. Trends Pharmacol Sci. 2020 Jan;41(1):4-12. doi: 10.1016/j.tips.2019.11.003. Epub 2019 Dec 10. PMID 31836191